CLINICAL TRIAL: NCT03779594
Title: Acetazolamide for Treating NPH in Shunt-candidates Patients: an Open Label Feasibility Trial
Brief Title: Acetazolamide for Treating NPH in Shunt-candidates Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0597-18
Record Dates: First submitted 2018-12-10; First posted 2018-12-19 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Normal Pressure Hydrocephalus
Keywords: NPH; Acetazolamide
MeSH Terms: conditions — Hydrocephalus, Normal Pressure | interventions — Acetazolamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- treatment group (Experimental): patients who met the inclusion criteria will be allocated to the treatment group, and will receive acetazolamide from time of diagnosis until shunt surgery (2-6 weeks).
  Interventions: Drug: Acetazolamide

INTERVENTIONS:
Drug: Acetazolamide — Patients will be assign and treated by acetazolamide from time of allocation until surgery (2-6 weeks after treatment initiation). The maximal dose of acetazolamide will be the same dose used to treat glaucoma, considering similarity of patients' characteristics, such as age and polypharmacy. We will start at a low dose of 250 mg once a day, and increase it slowly to a maximal dose of 500 mg twice a day. Dose will be individualized according to side-effects and tolerability. Renal and liver function tests will be performed before initiation of treatment, and will be examined again two weeks after treatment had begun.
  Other Names: Diamox

SUMMARY:
Normal pressure hydrocephalus (NPH) consists of a triad of gait disturbance, cognitive deterioration, and urinary incontinence and is characterized by enlarged cerebral ventricles. Current treatment recommendations are based on surgical diversion of Cerebrospinal fluid (CSF), by a ventriculoperitoneal shunt. When patients are appropriately selected, shunting for NPH has a sustained effect in one-half to two-thirds of patients with a reasonable complication rate. However, evidence regarding the efficacy of shunt surgery consists largely of observational studies with relatively short-term follow-up.

With regards to the adverse effects of shunting, even though decreased substantially in recent years, shunt complications are still common. Recent studies report ten to twenty-two percent of serious adverse effects following shunt surgery, mainly subdural hematoma (SDH) requiring surgery, infection, and cerebral infarction or hemorrhage. Most complication occur in the first year after the procedure. Many others suffer from adverse events that considered non-serious, such as postural headache and asymptomatic SDH.

Since shunt complications are common and potentially severe, there is a need for a better way to identify those patients that will likely benefit from shunting, and find alternative treatments for those unwilling or unable to withstand surgery.

Acetazolamide has been shown to reduce the production of CSF in clinical cases of raised intracranial pressure. It is considered the drug of choice for the treatment of idiopathic intracranial hypertension (pseudotumor cerebri). Intuitively, acetazolamide can be effective for the treatment of NPH by reducing the volume of CSF in the brain, and serve as a medical alternative to shunting. Few case reports and small series demonstrated improvement in MRI abnormalities in NPH-patients after administrating the medication.

This open-label study will examine the feasibility and effectiveness of acetazolamide in NPH-diagnosed patients who are shunt-candidates. Patients will be treated from time of diagnosis, and gait and cognition will be evaluated after 2-6 weeks. This trial would possibly pave the way to a larger randomized placebo-controlled trials, and perhaps offer a medical alternative to surgery for elderly patients and for patients for which operation is contraindicated.

ELIGIBILITY:
Inclusion Criteria:

Included will be subjects with a probable diagnosis of NPH. The diagnosis will be based primarily on presence of gait impairment plus at least one other impairment in urinary symptoms, cognition impairment or both.

1. Are 50 years old or older.
2. Patients who meet the criteria for NPH based on:

   * A typical personal history.
   * A typical brain imaging on head CT or MRI.
   * Normal lumbar puncture findings excluding other conditions.
   * Exclusion of other more likely diagnosis.
3. Patients who underwent large-volume spinal tap and subsequently improved clinically by at least 10% in gait function or cognition.

Exclusion Criteria:

* Cirrhosis or marked liver disease or dysfunction.
* Severe renal disease or dysfunction.
* Acidosis.
* Hypersensitivity to acetazolamide, sulfonamides, or any component of the formulation.
* Decreased sodium and/or potassium levels.
* Adrenocortical insufficiency.
* Patients with cognitive impairment who will not be able to give informed consent.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2018-12 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Gait | Baseline, week 4
  Change from Baseline gait will be evaluated by the neurosurgery department's physiotherapist, using the timed-up-and-go (TUG) test (measured in seconds, higher values represent a worse outcome).
  Patients will be evaluated at baseline (before treatment is started) and again before surgery (4 weeks later).
Change from Baseline Balance | Baseline, week 4
  Change from Baseline balance will be evaluated by the neurosurgery department's physiotherapist, using the TINETTI balance assessment score. (0-28 scale, higher values represent a better outcome).
  Patients will be evaluated at baseline (before treatment is started) and again before surgery (4 weeks later).

SECONDARY OUTCOMES:
Change from Baseline concentration function | Baseline, week 4
  concentration function will be evaluated by the neurosurgery department's neuropsychologist using the color trial test (seconds, higher values represent a worse outcome).
  Patients will be evaluated at baseline (before treatment is started) and again before surgery (4 weeks later).
Change from Baseline visuospatial function | Baseline, week 4
  visuospatial function will be evaluated by the neurosurgery department's neuropsychologist using the clock drawing test (0-10 scale, higher values represent a better outcome).
  Patients will be evaluated at baseline (before treatment is started) and again before surgery (4 weeks later).
Change from Baseline verbal fluency | Baseline, week 4
  verbal fluency will be evaluated by the neurosurgery department's neuropsychologist using the verbal fluency test (Controlled Oral Word Association Test, number of words in one minute, higher values represent a better outcome).
  Patients will be evaluated at baseline (before treatment is started) and again before surgery (4 weeks later).

OTHER OUTCOMES:
adverse effects | week 2-6
  All adverse effects that may be attributed to the treatment will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Yosi Laviv, MD, Principal Investigator — Rabin Medical Center
Locations (1):
- Rabin Medical Center, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jaraj D, Rabiei K, Marlow T, Jensen C, Skoog I, Wikkelso C. Prevalence of idiopathic normal-pressure hydrocephalus. Neurology. 2014 Apr 22;82(16):1449-54. doi: 10.1212/WNL.0000000000000342. Epub 2014 Mar 28. PMID 24682964
- [Background] Kuriyama N, Miyajima M, Nakajima M, Kurosawa M, Fukushima W, Watanabe Y, Ozaki E, Hirota Y, Tamakoshi A, Mori E, Kato T, Tokuda T, Urae A, Arai H. Nationwide hospital-based survey of idiopathic normal pressure hydrocephalus in Japan: Epidemiological and clinical characteristics. Brain Behav. 2017 Jan 27;7(3):e00635. doi: 10.1002/brb3.635. eCollection 2017 Mar. PMID 28293475
- [Background] Halperin JJ, Kurlan R, Schwalb JM, Cusimano MD, Gronseth G, Gloss D. Practice guideline: Idiopathic normal pressure hydrocephalus: Response to shunting and predictors of response: Report of the Guideline Development, Dissemination, and Implementation Subcommittee of the American Academy of Neurology. Neurology. 2015 Dec 8;85(23):2063-71. doi: 10.1212/WNL.0000000000002193. PMID 26644048
- [Background] Klassen BT, Ahlskog JE. Normal pressure hydrocephalus: how often does the diagnosis hold water? Neurology. 2011 Sep 20;77(12):1119-25. doi: 10.1212/WNL.0b013e31822f02f5. Epub 2011 Aug 17. PMID 21849644
- [Background] Esmonde T, Cooke S. Shunting for normal pressure hydrocephalus (NPH). Cochrane Database Syst Rev. 2002;2002(3):CD003157. doi: 10.1002/14651858.CD003157. PMID 12137677
- [Background] Tisell M, Tullberg M, Hellstrom P, Edsbagge M, Hogfeldt M, Wikkelso C. Shunt surgery in patients with hydrocephalus and white matter changes. J Neurosurg. 2011 May;114(5):1432-8. doi: 10.3171/2010.11.JNS10967. Epub 2011 Jan 14. PMID 21235310
- [Background] Kazui H, Miyajima M, Mori E, Ishikawa M; SINPHONI-2 Investigators. Lumboperitoneal shunt surgery for idiopathic normal pressure hydrocephalus (SINPHONI-2): an open-label randomised trial. Lancet Neurol. 2015 Jun;14(6):585-94. doi: 10.1016/S1474-4422(15)00046-0. Epub 2015 Apr 28. PMID 25934242
- [Background] Toma AK, Papadopoulos MC, Stapleton S, Kitchen ND, Watkins LD. Systematic review of the outcome of shunt surgery in idiopathic normal-pressure hydrocephalus. Acta Neurochir (Wien). 2013 Oct;155(10):1977-80. doi: 10.1007/s00701-013-1835-5. Epub 2013 Aug 23. PMID 23975646
- [Background] ten Hove MW, Friedman DI, Patel AD, Irrcher I, Wall M, McDermott MP; NORDIC Idiopathic Intracranial Hypertension Study Group. Safety and Tolerability of Acetazolamide in the Idiopathic Intracranial Hypertension Treatment Trial. J Neuroophthalmol. 2016 Mar;36(1):13-9. doi: 10.1097/WNO.0000000000000322. PMID 26587993
- [Background] Alperin N, Oliu CJ, Bagci AM, Lee SH, Kovanlikaya I, Adams D, Katzen H, Ivkovic M, Heier L, Relkin N. Low-dose acetazolamide reverses periventricular white matter hyperintensities in iNPH. Neurology. 2014 Apr 15;82(15):1347-51. doi: 10.1212/WNL.0000000000000313. Epub 2014 Mar 14. PMID 24634454
- [Background] Ivkovic M, Reiss-Zimmermann M, Katzen H, Preuss M, Kovanlikaya I, Heier L, Alperin N, Hoffmann KT, Relkin N. MRI assessment of the effects of acetazolamide and external lumbar drainage in idiopathic normal pressure hydrocephalus. Fluids Barriers CNS. 2015 Apr 2;12:9. doi: 10.1186/s12987-015-0004-z. PMID 25928394